CLINICAL TRIAL: NCT06544018
Title: Identification of Circadian Rhythm Deregulation in Patients With Cryopyrin-associated Periodic Syndrome (CAPS)
Brief Title: Circadian Rhythm Deregulation in Patients With CAPS
Acronym: ICARUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_0417; 2023-A01088-37 (Other: ID-RCB)
Record Dates: First submitted 2024-05-07; First posted 2024-08-09 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cryopyrin Associated Periodic Syndrome; Familial Cold Urticaria; Muckle-Wells Syndrome; CINCA Syndrome
Keywords: Circadian clock; cryopyrin-associated periodic syndrome; familial cold urticaria; muckle-wells syndrome; melatonin
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, interventional, comparative, open-label, controlled study with 2 parallel arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with cryopyrin-associated periodic syndrome (CAPS) (Active Comparator): Confirmed by genetic analysis of NLRP3
  Interventions: Genetic: Genetic analysis of NLRP3; Device: Circadian rhythm measurement; Biological: Saliva sampling; Other: Questionnaire; Other: AIDAI score; Biological: Blood sampling
- Control group (Placebo Comparator): Healthy participant (absence of CAPS, verified by NLRP3 gene analysis) living in the same household as a CAPS participant included in the protocol
  Interventions: Genetic: Genetic analysis of NLRP3; Device: Circadian rhythm measurement; Biological: Saliva sampling; Other: Questionnaire; Biological: Blood sampling

INTERVENTIONS:
Genetic: Genetic analysis of NLRP3 — Blood test for genetic analysis of NLRP3
Device: Circadian rhythm measurement — Wear a Withings Pulse HR (heart rate) actigraphic watch 24 hours a day for 1 month to define circadian rhythm
Biological: Saliva sampling — Saliva sampling for salivary melatonin determination
Other: Questionnaire — Questionnaire to determine chronotype
Other: AIDAI score — Disease activity score using AIDAI score (only for patients in the CAPS group) AIDAI : AUTO-INFLAMMATORY DISEASE ACTIVITY INDEX
  Arms: Patients with cryopyrin-associated periodic syndrome (CAPS)
Biological: Blood sampling — 1. Inflammatory cytokines measurement : IL1-beta (Interleukin-1) and IL-18.
  2. Molecular characterization of circadian clock signaling pathways

SUMMARY:
Circadian rhythms are characterized by the physiology's adaptation to the alternation of day and night, enabling to adapt to the environment. These rhythms are generated by a molecular clock within each cell. At the molecular level, the circadian clock is based on a complex system of cell-autonomous transcription loops. These exert positive and negative feedback on themselves, generating cyclic transcriptional activity.

* In the main loop, the BMAL1 transcription factor links with CLOCK or NPAS2 ( (Neuronal PAS Domain Protein 2) to activate transcription of per1,2 and 3 and cryptochrome (cry1 and cry2), which in turn repress BMAL1/CLOCK1 transcriptional activity.. The BMAL1/CLOCK complex also activates transcription of numerous target genes (per and cry, Rev-erb, etc.)..
* other secondary loops refine the function of the first.

Recent studies suggest that many aspects of innate immunity are controlled by circadian rhythm through inhibition of NLRP3 inflammasome activation. Nevertheless, the regulation of the NLRP3 inflammasome by the circadian clock has yet to be elucidated. Inflammasomes are molecular platforms that control caspase-1 activation and consequently the maturation of precursors of (interleukine) IL-1β, pro-IL-18, a pro-inflammatory cytokine. Since its discovery, its functions have been widely characterized as part of the innate immune response as a sensor of pathogens and danger signals (extracellular ATP (Adenosine triphosphate), atmospheric pollutants). NLRP3 (nucleotide-binding domain LRR (leucin-rich repeat ) and pyrin-containing receptor 3) has been described for its genetic association with dominant monogenic hereditary syndromes characterized by recurrent systemic inflammatory episodes in the absence of any infection or autoimmune disease, known as CAPS (cryopyrin-associated periodic syndrome) or cryopyrinopathies which is a continuum of diseases ranging from a moderate to the most severe form of the syndrome: familial cold urticaria syndrome, Muckle-Wells syndrome (MWS), and CINCA/NOMID syndrome.

Interestingly, patients with Muckle-Wells syndrome show a circadian pattern of symptoms, with a recurrent, predominantly vesperal fever peak lasting a few hours, and extreme fatigue on a daily basis. However, a molecular link between the circadian clock and CAPS pathology remains to be determined.

The aim of this protocol is to identify circadian rhythm dysregulation in patients with CAPS confirmed by genetic analysis of NLRP3, to demonstrate a link between circadian clock and CAPS syndrome, and to identify circadian clock regulatory pathways.

ELIGIBILITY:
---Inclusion Criteria:

Patient with CAPS group :

* Patients aged 6 and over
* Participant with CAPS confirmed by NLRP3 genetic analysis
* Weight greater than or equal to 25 Kg
* Parents/guardians who have been informed of the study and have signed a consent form.
* Patient affiliated to a social security scheme

Control group (healthy participant):

* Participant aged 6 and over
* Weight greater than or equal to 25 Kg
* Participant living in the same household as a subject with CAPS genetically confirmed by NLRP3 analysis and included in the protocol
* Participant with no CAPS (a priori) who consents to NLRP3 genetic analysis
* Parents/guardians who have been informed of the study and have signed a consent form.
* Participant who has been informed of the study and has agreed to take part
* Participant affiliated to a social security scheme

  * Exclusion Criteria :

Patient with CAPS group :

* Patients with chronic sleep disorders (narcolepsy, hypersomnia) requiring medication (sleeping pills, melatonin).
* Patients with sleep apnea syndrome
* Patients working regular night shifts or alternating day and night shifts
* Pregnant or breast-feeding women
* Parents with an infant under 6 months of age
* Patient participating in another interventional drug study
* Deprivation of civil rights (curators, guardianship, safeguard of justice)

Control group (healthy participant):

* Participants with a chronic illness (ALD beneficiaries)
* Participants with chronic sleep disorders (narcolepsy, hypersomnia) requiring medication (sleeping pills, melatonin)
* Participants working regular night shifts or alternating day and night shifts
* Pregnant or breast-feeding women
* Parents with an infant under 6 months of age
* Participant participating in another interventional drug study
* Deprivation of civil rights (curators, guardianship, safeguard of justice)

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Description of circadian rhythm deregulation in patients with cryopyrinopathy (CAPS) whose diagnosis was confirmed by genetic analysis of NLRP3, | 6 months after inclusion
  Concentration of the peak secretion of melatonin in both arms
Description of circadian rhythm deregulation in patients with cryopyrinopathy (CAPS) whose diagnosis was confirmed by genetic analysis of NLRP3, | 12 months after inclusion
  Concentration of the peak secretion of melatonin in both arms
Description of circadian rhythm deregulation in patients with cryopyrinopathy (CAPS) whose diagnosis was confirmed by genetic analysis of NLRP3, | 6 months after inclusion
  time of the peak secretion of melatonin in both arms
Description of circadian rhythm deregulation in patients with cryopyrinopathy (CAPS) whose diagnosis was confirmed by genetic analysis of NLRP3, | 12 months after inclusion
  time of the peak secretion of melatonin in both arms

SECONDARY OUTCOMES:
Difference in circadian clock biomarkers between patients and control participants for Circadian Rhythm Characteristics. | 6 th month
  Determination of circadian rhythms : amplitude in both arms
Difference in circadian clock biomarkers between patients and control participants for Circadian Rhythm Characteristics. | 6 th month
  Determination of circadian rhythms : period in both arms
Difference in circadian clock biomarkers between patients and control participants for Circadian Rhythm Characteristics. | 6 th month
  Determination of circadian rhythms : phase in both arms
Chronotype determination | 6 th month
  Number of patients in each chronotype for the 2 arms based on the specific questionnaire in both arm
sleep duration | 6 th month
  sleep duration in both arms
number of steps | 6 th month
  Daily activity in both arms
Comparison of inflammatory state | 6 months after inclusion
  basal levels of IL1β in patient monocytes in both arms
Comparison of inflammatory state | 12 months after inclusion
  basal levels of IL1β in patient monocytes in both arms
Comparison of inflammatory state | 6 months after inclusion
  basal levels of IL18 in patient monocytes in both arms
Comparison of inflammatory state | 12 months after inclusion
  basal levels of IL18 in patient monocytes in both arms
Disease activity measurement | 6 months after inclusion
  Number of patient with active disease ie AIDAI (AUTO-INFLAMMATORY DISEASE ACTIVITY INDEX) score >9 in CAPS patient arm
Disease activity measurement | 12 months after inclusion
  Number of patient with active disease ie AIDAI (AUTO-INFLAMMATORY DISEASE ACTIVITY INDEX) score >9 in CAPS patient arm
presence or absence of an abnormality in the NLRP3 signalling pathway in CAPS arm compared control arm | 6 months after inclusion
  Biochemical characterization of the NLRP3 inflammasome protein regulatory pathway in both arms
presence or absence of an abnormality in the NLRP3 signalling pathway in CAPS arm compared to control arm | 12 months after inclusion
  Biochemical characterization of the NLRP3 inflammasome protein regulatory pathway in both arms
presence or absence of ASC inflammasome protein regulatory pathway in CAPs arm compared to control arm | 6 months after inclusion
  Biochemical characterization of the ASC inflammasome protein regulatory pathway in both arms
presence or absence of ASC inflammasome protein regulatory pathway in CAPS arm compared to control arm | 12 months after inclusion
  Biochemical characterization of the ASC inflammasome protein regulatory pathway in both arms
presence or absence of the CASPASE-1 inflammasome protein regulatory pathway in CAPS arm compared to control arm | 6 months after inclusion
  Biochemical characterization of the CASPASE-1 inflammasome protein regulatory pathway in both arms
presence or absence of the CASPASE-1 inflammasome protein regulatory pathway in CAPS arm compared to control arm | 12 months after inclusion
  Biochemical characterization of the CASPASE-1 inflammasome protein regulatory pathway in both arms
presence or absence of REV-ERBα inflammasome protein regulatory pathway in CAPS arm compared to control arm | 6 months after inclusion
  Biochemical characterization of the REV-ERBα inflammasome protein regulatory pathway in both arms
presence or absence of REV-ERBα inflammasome protein regulatory pathway in CAPS arm compared to control arm | 12 months after inclusion
  Biochemical characterization of the REV-ERBα inflammasome protein regulatory pathway in both arms

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hôpital Femme-Mère-Enfant (HCL), Bron
  - Hôpital Claude Huriez (CHU de Lille), Lille
  - Hôpital de la Croix-Rousse (HCL), Lyon
  - Hôpital Edouard Herriot (HCL), Lyon
  - Hôpital Tenon (AP-HP), Paris
  - Hôpital Kremlin-Bicêtre (AP-HP), Paris

IPD SHARING:
Plan to Share IPD: No